CLINICAL TRIAL: NCT02231164
Title: Multicentre, Randomised, Double-blind, Phase III Trial to Investigate the Efficacy and Safety of Oral Nintedanib Plus Docetaxel Therapy Compared to Placebo Plus Docetaxel Therapy in Patients With Stage IIIB/IV or Recurrent, Adenocarcinoma Subtype Non-small Cell Lung Cancer After Failure of First Line Chemotherapy
Brief Title: LUME-Columbus: Nintedanib Plus Docetaxel in Advanced Non-small Cell Lung Cancer With Translational Research
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1199.128
Record Dates: First submitted 2014-09-02; First posted 2014-09-04 (Estimated); Results first posted 2017-02-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-01

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Docetaxel; nintedanib

ARMS (2):
- Docetaxel and placebo (Placebo Comparator): patients to receive backbone chemotherapy and placebo
  Interventions: Drug: docetaxel; Drug: placebo
- Docetaxel and Nintedanib (Experimental): patients to receive backbone chemotherapy and nintedanib
  Interventions: Drug: docetaxel; Drug: nintedanib

INTERVENTIONS:
Drug: docetaxel — intravenous chemotherapy drug
  Arms: Docetaxel and Nintedanib
Drug: docetaxel — intravenous chemotherapy drug
  Arms: Docetaxel and placebo
Drug: placebo — oral placebo
  Arms: Docetaxel and placebo
Drug: nintedanib — oral experimental therapy
  Arms: Docetaxel and Nintedanib

SUMMARY:
The present trial will investigate the efficacy and safety of nintedanib in combination with docetaxel as compared to placebo in combination with docetaxel in patients with stage IIIB/IV or recurrent NSCLC of adenocarcinoma histology after failure of first-line platinum-based chemotherapy.

ELIGIBILITY:
Inclusion criteria:

* Male or female patients of at least 18 years of age
* Histologically confirmed, adenocarcinoma of the lung, after failure of first line platinum-based chemotherapy.

Exclusion criteria:

* More than one prior line of chemotherapy (i.e., 2nd or 3rd line chemotherapy) for advanced and/or metastatic (stage III B or IV NSCLC) or recurrent disease.
* Patients known to be positive for activating Epidermal Growth Factor Receptor (EGFR) mutation or anaplastic lymphoma kinase (ALK) translocation
* Previous therapy with other vascular endothelial growth factor (VEGF) or VEGFR inhibitors (other than bevacizumab) or docetaxel for the treatment of NSCLC at any time
* Prior monotherapy with an EGFR inhibitor except as maintenance therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-10-14 (Actual); Primary Completion 2015-12-24 (Actual); Study Completion 2015-12-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (13):
- United States (9):
  - 1199.128.10032 Boehringer Ingelheim Investigational Site, Chandler, Arizona
  - 1199.128.10041 Boehringer Ingelheim Investigational Site, Fayetteville, Arkansas
  - 1199.128.10010 Boehringer Ingelheim Investigational Site, Highland, California
  - 1199.128.10044 Boehringer Ingelheim Investigational Site, Rancho Mirage, California
  - 1199.128.10080 Boehringer Ingelheim Investigational Site, Paducah, Kentucky
  - 1199.128.10016 Boehringer Ingelheim Investigational Site, Farmington, New Mexico
  - 1199.128.10013 Boehringer Ingelheim Investigational Site, Minot, North Dakota
  - 1199.128.10077 Boehringer Ingelheim Investigational Site, Blacksburg, Virginia
  - 1199.128.10011 Boehringer Ingelheim Investigational Site, Kennewick, Washington
- Georgia (3):
  - 1199.128.64006 Boehringer Ingelheim Investigational Site, Batumi
  - 1199.128.64001 Boehringer Ingelheim Investigational Site, Tbilisi
  - 1199.128.64002 Boehringer Ingelheim Investigational Site, Tbilisi
- 1199.128.66004 Boehringer Ingelheim Investigational Site, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo soft gelatin capsule matching that of nintedanib twice daily on Day 2 to 21 of each 21-day treatment course administered orally plus docetaxel 75 mg/m^2 on Day 1 of each 21-day treatment course administered via intravenous infusion. If required the dose of placebo could be reduced to 150 mg twice daily (b.i.d.) or 100 mg b.i.d and one dose reduction was permitted for docetaxel (according to the protocol-defined dose-reduction scheme). No dose increase was allowed after a dose reduction.
- Nintedanib: Nintedanib 200 mg twice daily (b.i.d.) on Day 2 to 21 of each 21-day treatment course administered orally in the form of a soft gelatin capsule plus docetaxel 75 mg/m^2 on Day 1 of each 21-day treatment course administered via intravenous infusion. If required the dose of nintedanib, could be reduced to 150 mg b.i.d. or 100 mg b.i.d. and one dose reduction was permitted for Docetaxel (according to the protocol-defined dose-reduction scheme). No dose increase was allowed after a dose reduction.
Period: Overall Study
Arm/Group | Placebo | Nintedanib
Started | 6 | 6
Completed | 0 | 0
Not Completed | 6 | 6
Not completed — Adverse Event | 1 | 1
Not completed — Lack of Efficacy | 4 | 3
Not completed — Withdrawal by Subject | 1 | 2

BASELINE CHARACTERISTICS:
Population: Randomised Set: The randomised set included all randomised patients.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Nintedanib | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.7 (12.2) | 63.3 (8.3) | 61.5 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 5 | 4 | 9

OUTCOME MEASURES:

1. Primary Outcome: Disease Control According to Response Evaluation Criteria in Solid Tumours (RECIST), Version 1.1
Description: This outcome measure presents the number of patients with disease control according to RECIST, version 1.1, defined as number of patients with Complete response, partial response or stable disease.
Time Frame: Up to 6 months.
Population: Randomised Set: The randomised set included all randomised patients.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Nintedanib
Number analyzed (Participants) | 6 | 6
Percentage of participants
  Yes | 66.7 | 50.0
  No | 33.3 | 50.0

ADVERSE EVENTS:
Time Frame: From first drug administration until 28 days after last drug administration, up to 7 months.
Arm/Group | Placebo | Nintedanib
Serious Adverse Events (participants affected / at risk) | 3/6 | 3/6
Other Adverse Events (participants affected / at risk) | 5/6 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=6) | Nintedanib (N=6)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Clostridium difficile infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 1
Sepsis (Infections and infestations) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Metastases to skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Orthostatic hypotension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=6) | Nintedanib (N=6)
Anaemia (Blood and lymphatic system disorders) | 2 | 0
Leukopenia (Blood and lymphatic system disorders) | 2 | 1
Neutropenia (Blood and lymphatic system disorders) | 2 | 3
Lacrimation increased (Eye disorders) | 1 | 1
Visual impairment (Eye disorders) | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 3 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 4
Dry mouth (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1
Frequent bowel movements (Gastrointestinal disorders) | 0 | 1
Glossodynia (Gastrointestinal disorders) | 1 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 5
Oral pain (Gastrointestinal disorders) | 0 | 2
Stomatitis (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 5
Chest pain (General disorders) | 0 | 1
Chills (General disorders) | 1 | 1
Facial pain (General disorders) | 0 | 1
Fatigue (General disorders) | 4 | 3
Mucosal inflammation (General disorders) | 1 | 1
Oedema peripheral (General disorders) | 1 | 0
Pain (General disorders) | 2 | 1
Polyp (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Allergy to arthropod sting (Immune system disorders) | 0 | 1
Seasonal allergy (Immune system disorders) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Breath sounds abnormal (Investigations) | 0 | 1
Weight decreased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 2 | 4
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Dysgeusia (Nervous system disorders) | 1 | 2
Headache (Nervous system disorders) | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 1 | 3
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 2
Mood altered (Psychiatric disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 1 | 1
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 2
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 | 1
Nail ridging (Skin and subcutaneous tissue disorders) | 1 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 2
Phlebitis (Vascular disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
The sponsor cancelled this trial prematurely. Thus, enrollment for 1199.128 was significantly less than what was planned (800 planned vs. 12 entered). Therefore, the objectives of this study could not be fully assessed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.